CLINICAL TRIAL: NCT02456948
Title: A Double-blind, Placebo-controlled, Randomized, Multicenter Proof-of-principle Trial of Adjunctive Minocycline for Patients With Unipolar Major Depressive Disorder (MDD)
Brief Title: Adjunct Minocyline in Treatment-resistant Depression
Acronym: Mino-TRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Isabella Heuser, MD, PhD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01EE1401F
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
Keywords: treatment resistant depression; inflammation; microglia; minocycline
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Inflammation; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): Minocycline and standard antidepressant treatment
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Placebo and standard antidepressant treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — 6 weeks 200mg/day Minocycline add-on
  Other Names: Solodyn; Minocin
  Arms: Minocycline
Drug: Placebo — 6 weeks Placebo add-on
  Other Names: Sugar pills, mimics Minocycline tablet
  Arms: Placebo

SUMMARY:
This study examines the antidepressant efficacy of minocycline as an adjunct to an antidepressant standard treatment (AD-ST), for patients with unipolar major depressive disorder (MDD).

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, multicenter proof-of-principle trial of adjunctive minocycline for patients with unipolar major depressive disorder (MDD). The study tests the antidepressant efficacy of minocycline as an adjunct to an antidepressant standard treatment (AD-ST), for patients with unipolar major depressive disorder (MDD). The respective AD, for which non-response has been documented, must be on a stable regimen for at least 14 days prior to inclusion. AD-ST will then be continued throughout the trial. Trial medication is adjunct oral minocycline 200 mg/day or placebo. Response to treatment will be measured via the Montgomery-Asberg Depression Rating Scale (MADRS). The total study duration for each patient will be 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* male or female
* between age 18 and 75
* BMI between 18 and 40 inclusive
* Non-lactating, non-pregnant females of child-bearing potential must be willing to use an effective contraceptive method
* All participants must fulfil diagnostic criteria of moderate or severe MDD according to the DSM-5.
* HAMD-17 score of at least 16 points at baseline and a
* CGI-S score of at least 4.
* AD-ST must have been administered at a sufficient dose for at least 6 weeks in the current episode and at a
* stable regimen for at least 14 days prior to baseline.
* Dose and duration of AD-ST must be verifiable

Exclusion Criteria:

* prevalence of neurodegenerative disorder
* prevalence of any neurological disorder that caused the depressive symptoms
* prevalence of any severe, unstable general medical condition, including chronic inflammatory disease such as rheumatoid arthritis or inflammatory bowel disease
* prevalence of any other psychiatric disorder that better explains the presence of depressive symptoms
* Improvement by more than 50% in HAMD-17 score during the last 14 days prior to baseline
* pregnant or nursing women will not be allowed.
* substance or alcohol abuse within past 6 months or positive urine drug screening
* abnormal thyroid function (euthyroid at presentation), liver or kidney dysfunction
* history of autoimmune disease (except Hashimotos thyroiditis)
* clinically significant laboratory abnormalities (outside normal ranges)
* current medication with anti-inflammatory substances (NSAIDs, corticosteroids)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Response as per MADRS (Montgomery-Åsberg Depression Rating Scale) | 6 weeks

SECONDARY OUTCOMES:
Remission as per MADRS (Montgomery-Åsberg Depression Rating Scale) | 6 weeks
HAM-D-17-Scale (17-item Hamilton Depression Rating Scale) | 6 weeks
BDI-Scale (Beck Depression Inventory, Self Rating Scale) | 6 weeks
CGI-Scale (Clinical Global Impressions Scale) | 6 weeks
SCL-90-R (Symptom Checklist 90-R, Self Rating Scale) | 6 weeks
Transcriptomic changes in patient-specific peripheral blood-derived monocytic cells | 6 weeks
Protein levels of various inflammation-associated markers in patient sera | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Heuser, MD, PhD, Principal Investigator — Chair: Department of Psychiatry Charité - Campus Benjamn
Locations (9):
- Germany (9):
  - Heidelberg University Hospital, Department of Psychiatry, Heidelberg, Baden-Wurttemberg
  - Department of Psychiatry, Universitiy Hospital, Erlangen, Bavaria
  - Department of Psychiatry, LMU Munich, Munich, Bavaria
  - Max Planck Institute of Psychiatry, Munich, Bavaria
  - Department of Psychiatry, Universitiy Hospital, Regensburg, Bavaria
  - Department of Psychiatry, University Medical Center Göttingen, Göttingen, Lower Saxony
  - Department of Psychiatry, Psychotherapy and Psychosomatics, University Hospital RWTH Aachen, Aachen
  - Department of Psychiatry, Charité - Campus Benjamin Franklin, Berlin
  - Dept. of Psychiatry, Psychosomatic Medicine and Psychotherapy, University Hospital Frankfurt, Frankfurt

IPD SHARING:
Plan to Share IPD: No